CLINICAL TRIAL: NCT06808464
Title: Evaluation of Autonomic Activity in REM Sleep by a New Marker of Cardiac Variability in Subjects With Severe Obstructive Sleep Apnea Hypopnea Syndrome
Brief Title: New Approach in the Study of the Autonomic Nervous System Through Cardiac Variability in Sleep Apnea Syndrome.
Acronym: HRVSAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_0403; 2022-A01069-34 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea hypopnea syndrome; Autonomic nervous system; Cardiac variability; Automatic detection; Machine Learning
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Arm "experimental" consists in questioners and polysomnography on patients with severe sleep apnea
- Control group: Arm "control" consists in questioners and polysomnography on healthy subjects

SUMMARY:
The main objective of this study is to compare the different variations of the cardiac variability index measured thanks to the technique developed by the CIC-IT between subjects with severe SAS and healthy subjects with sleep pathology.

In a first step, these two groups will be compared in REM sleep phase because it is the period during which the risk of sleep apnea syndrome is the highest. In a second step, the same methodology will be applied for the other sleep phases and correlations will be established with the other markers of cardiac variability (HRV) already known. This will allow to validate a reliable method of screening for SAS that is more accessible in ambulatory settings by means of a machine learning system based on artificial intelligence

ELIGIBILITY:
Inclusion Criteria:

* Group healthy subjects - 1): absence of sleep disorder referenced in the ICSD-3.

  * Epworth Sleep Scale < 11
  * Pittsburgh Quality Sleep Index < 6
  * Berlin Questionnaire: < 2 positive categories
  * STOP BANG <3
  * HADS normal
  * No RLS
* Group 2 (subjects with severe SAS - 2): AHI > 30/h obstructive

Exclusion Criteria:

Non-inclusion criteria:

* Cardiac rhythm disorder
* Neurological or psychiatric pathology impacting on ANS
* Control group (healthy subjects - 1)

  * Complaint of sleep disorder
  * Known sleep disorder
* Experimental group (subjects with severe SAS - 2):

  o Associated sleep pathology at diagnosis of severe SAS
* Administrative reasons:

  * Unable to receive informed information,
  * Unable to participate in the entire study
  * Lack of social security coverage
  * Refusal to sign consent Exclusion criteria
* Control group (healthy subjects - 1):

  * Sleep pathology detected by polysomnography
  * Total sleep time less than 4 hours
  * Recording technically not usable

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruitment of patients after the diagnosis of severe SAS in the services of the University Hospital of Lille. The healthy subjects will be recruited through an advertisement in the general medicine networks of the Hauts de France region.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Ability of the high frequency variability index (HFVI) measured in REM sleep phase to differentiate subjects with severe SAS and healthy subjects with sleep pathology | Baseline (The day of the polysomnography )

SECONDARY OUTCOMES:
Mean value of the IVHF in the other sleep stages (N1, N2 and N3) | Baseline (The day of the polysomnography )
  Variations of the IVHF between subjects with severe SAS and healthy subjects for the other sleep stages
Mean value of other VFC variables in the different sleep stages (REM, N1, N2 and N3) | Baseline (The day of the polysomnography )
  Variations of the other markers of cardiac variability between subjects with severe SAS and healthy subjects for all sleep phases
Total score and sub-score of the SCOPA-AUT questionnaire (between 0-69), with the possibility of analysis of the different sub-scores. | Baseline (The day of the polysomnography )
  Variation of other nervous system components by standardized questionnaire between a group with severe SAS and a group of control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DERAMBURE, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service de Neurophysiologie - unité de médecine du Sommeil - CHU Lille, Lille, France